CLINICAL TRIAL: NCT02353052
Title: Prospective Cohort Study of the Clinical Applications for the Pathologic Type, Staging, and Grading of Primary Gastrointestinal Stromal Tumor
Brief Title: Prospective Cohort Study of the Clinical Applications for the Pathologic Type, Staging, and Grading of GIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiZhongshan
Record Dates: First submitted 2015-01-17; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: morphology standards
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — GIST paraffin specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treatment observation group: According to the morphological criteria, the NIH scheme, and the WHO standard, GIST patients are divided into two groups, benign group and malignant group. In fully informed of their illness, patients are free to choose the sequence treatments according to their own gene mutation status and economic conditions. Patients who choose postoperative Imatinib treatment are labeled treatment group.
  Interventions: Other: follow up
- Control observation group: According to the morphological criteria, the NIH scheme, and the WHO standard, GIST patients are divided into two groups, benign group and malignant group. In fully informed of their illness, patients are free to choose the sequence treatments according to their own gene mutation status and economic conditions. Patients who choose no Imatinib treatment are labeled observation group.
  Interventions: Other: follow up

INTERVENTIONS:
Other: follow up — The patients were followed up for 3 years about their survival conditions and tumor status (eg. recurrence and metastasis).

SUMMARY:
Evaluate the reliability of morphology standards for GIST pathologic type, staging and grading by retrospective analyzing clinical data; on this basis, establish a GIST standardized and individualized treatment mode to maximum benefit GIST patients, avoid under- and over-treatment.

DETAILED DESCRIPTION:
1. Retrospective analysis of GIST cases in the recent five years: the GIST clinical data of Fudan University Zhongshan Hospital from 2007 January to 2012 December were collected. By reviewing the HE slides, GIST was evaluated by 12 indicators, NIH scheme and WHO standard. Accomplish the gene sequencing of KIT, PDGFRA, B-raf, and SDH. Follow up the patients about their treatment and prognosis. Analyze and compare the advantages and disadvantages of the histomorphology indicators, NIH scheme, and WHO standard.
2. Organize the first prospective cohort study of GIST individualized treatment based on the histomorphology. Obtain the evidence of histological assessment for GIST by following up patients for 3 years.
3. Establish an evaluation criteria based on the morphology of GIST. Make objective evaluations about GIST tumor size, tumor location and gene mutation status in the prognosis estimate. Make rules to effectively guide individualized treatment of GIST.

ELIGIBILITY:
All patients pathologically diagnosed with GIST during the period from 2013 to 2015

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with GIST by pathology
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tumor recurrence | 3 years
Number of participants with tumor metastasis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yingyong Hou, Doctor, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China